CLINICAL TRIAL: NCT00545051
Title: A Randomized, Double-blind Study to Evaluate the Effect of Once Monthly Bonviva on Lumbar Bone Mineral Density in the Prevention of Glucocorticoid-induced Osteoporosis in Post-menopausal Women
Brief Title: A Study of Once Monthly Bonviva (Ibandronate) in Prevention of Glucocorticoid-Induced Osteoporosis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML20088
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ibandronate (Experimental): Participants received monthly oral ibandronate (150 milligrams [mg]) for 12 months.
  Interventions: Drug: ibandronate
- Placebo (Placebo Comparator): Participants received monthly oral placebo for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po monthly for 12 months
  Arms: Placebo
Drug: ibandronate — 150mg po monthly for 12 months
  Other Names: Bonviva/Boniva
  Arms: Ibandronate

SUMMARY:
This 2 arm study will investigate the efficacy and safety of Bonviva (150mg po monthly) in the prevention of glucocorticoid-induced osteoporosis in post-menopausal women. Patients will be randomized to receive either Bonviva 150mg po or placebo monthly, with vitamin D and calcium supplementation. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women, 50-85 years of age;
* any inflammatory rheumatoid disease including polymyalgia rheumatica;
* receiving treatment with 5-15 mg/day of prednisolone.

Exclusion Criteria:

* previous treatment with an iv bisphosphonate at any time;
* previous treatment with an oral bisphosphonate within the last 6 months, >1 month of treatment within last year, or >3 months of treatment within last 2 years;
* treatment with parathyroid hormone in last 2 years;
* inability to stand or sit in an upright position for at least 60 minutes;
* inability to swallow a tablet whole;
* history of major gastrointestinal disease.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Finland (10):
  - Hämeenlinna
  - Helsinki
  - Hyvinkää
  - Jyväskylä
  - Kuopio
  - Lahti
  - Oulu
  - Tampere
  - Turku
  - Vantaa

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibandronate: Participants received 150 milligram (mg) ibandronate tablet orally once a month for 12 months. Participants also received 1000 mg calcium and 800 International Units (IU) Vitamin D per day.
- Placebo: Participants received oral placebo tablet once a month for 12 months. Participants also received 1000 mg calcium and 800 IU Vitamin D per day.
Period: Overall Study
Arm/Group | Ibandronate | Placebo
Started | 68 | 72
Completed | 59 | 65
Not Completed | 9 | 7
Not completed — Adverse Event | 7 | 3
Not completed — Death | 1 | 0
Not completed — Violation of inclusion/exclusion | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Administrative reasons | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants randomized and who had at least one follow up efficacy data time point available.
Groups:
- Ibandronate: Participants received 150 mg ibandronate tablet orally once a month for 12 months. Participants also received 1000 mg calcium and 800 IU Vitamin D per day.
- Total: Total of all reporting groups
Arm/Group | Ibandronate | Placebo | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.90) | 63.2 (6.83) | 63.79 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 72 | 140
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Lumbar Spine Bone Mineral Density (BMD) at Month 12
Description: Lumbar spine BMD was measured at Baseline, and Months 6 and 12 using dual-energy x-ray absorptiometry (DXA). Percent change from Baseline to Month 12 was calculated using analysis of covariance.
Time Frame: Baseline and Month 12
Population: Intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 66 | 66
percent change in BMD | 3.2 (3.7) | -0.1 (3.0)
Statistical Analysis 1: Comparison: Ibandronate vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.25, 95% CI 2-sided [2.09 to 4.41]

2. Secondary Outcome: Percent Change From Baseline in Mean Lumbar Spine BMD at Month 6
Description: Lumbar spine BMD was measured at Baseline and Month 6 using DXA. Percent change from Baseline to Month 6 was calculated using analysis of covariance.
Time Frame: Baseline and Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 62 | 66
percent change in BMD | 2.6 (3.1) | 0.3 (2.8)
Statistical Analysis 1: Comparison: Ibandronate vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [1.22 to 3.23]

3. Secondary Outcome: Percent Change From Baseline in Mean Total Hip BMD at Month 6 and Month 12
Description: Left total hip BMD was measured by DXA at Baseline, and Months 6 and 12. If there was prosthesis of left hip, the measurement of right total hip BMD was done by DXA. Percent change from Baseline to Months 6 and 12 was calculated using analysis of (co)variance for repeated measurements.
Time Frame: Baseline and Months 6 and 12
Population: ITT population; number (n) equals (=) number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 66 | 66
percent change in BMD
  Month 6 (n=62,66) | 0.7 (1.9) | 0.0 (2.1)
  Month 12 (n=66,65) | 1.2 (2.2) | -0.7 (2.5)
Statistical Analysis 1: Comparison: Ibandronate vs Placebo; Month 6; Test type: Superiority or Other; p = 0.122, ANCOVA; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.15 to 1.25]
Statistical Analysis 2: Comparison: Ibandronate vs Placebo; Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [0.96 to 2.66]

4. Secondary Outcome: Percent Change From Baseline in Bone Turnover Markers at Month 1, Month 6 and Month 12
Description: Serum C-terminal Telopeptide of Type 1 Collagen (sCTX), Serum Procollagen Type 1 N-terminal Propeptide (P1NP) and Serum Bone Tartrate-resistant Acid Phosphatase Isoform 5b (TRACP) are measures of bone resorption and are measured as nanograms per milliliter (ng/mL). Percent change from Baseline to Months 1, 6 and 12 was calculated using analysis of covariance for repeated measurements.
Time Frame: Baseline and Months 1, 6 and 12
Population: ITT population; n=number of participants analyzed at the specified visit for the given parameter.
Measure: Mean (Standard Deviation); unit: percent change in bone turnover markers
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 68 | 68
percent change in bone turnover markers
  sCTX Month 1 (n=68,68) | -44.7 (36.5) | -3.8 (33.3)
  sCTX Month 6 (n=62,66) | -53.3 (24.3) | -3.5 (48.0)
  sCTX Month 12 (n=65,65) | -42.0 (27.9) | 11.6 (82.4)
  P1NP Month 1 (n=68,68) | -23.8 (17.2) | -2.3 (22.5)
  P1NP Month 6 (n=60,66) | -62.5 (16.3) | -3.7 (44.5)
  P1NP Month 12 (n=64,67) | -48.8 (37.2) | 12.5 (54.6)
  TRACP Month 1 (n=68,68) | -31.3 (12.0) | -7.3 (11.9)
  TRACP Month 6 (n=62,66) | -32.9 (14.8) | -7.1 (17.0)
  TRACP Month 12 (n=65,67) | -27.4 (16.5) | -6.3 (18.0)
Statistical Analysis 1: Comparison: Ibandronate vs Placebo; sCTX at Month 1; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Ibandronate vs Placebo; sCTX at Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Ibandronate vs Placebo; sCTX at Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Ibandronate vs Placebo; P1NP at Month 1; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Ibandronate vs Placebo; P1NP at Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Ibandronate vs Placebo; P1NP at Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Ibandronate vs Placebo; TRACP at Month 1; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Ibandronate vs Placebo; TRACP at Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Ibandronate vs Placebo; TRACP at Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Percentage of Participants Withdrawn Due to Worsening in BMD at 6 Months and/or Worsening in BMD at Least 7 Percent (%) at Any Site at 6 Months
Description: Worsening in BMD was defined as BMD T-score at any site less than or equal to (≤) - 2.5 standard deviations and/or worsening in BMD of at least 7% at any site.
Time Frame: Month 6
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 62 | 66
percentage of participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of randomization until 15 days after the end of study at 12 months.
Description: The safety population included all participants who had at least one dose of the trial medication, whether withdrawn prematurely or not, and at least one follow-up data point. Two participants received both treatments and were allocated to the ibandronate group for all assessments of safety.
Arm/Group | Ibandronate | Placebo
Serious Adverse Events (participants affected / at risk) | 10/70 | 6/70
Other Adverse Events (participants affected / at risk) | 19/70 | 26/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=70) | Placebo (N=70)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia due to gastrointestinal bleeding (Blood and lymphatic system disorders) | 1 | 0
Acute pancreatitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Acute pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Concussion (General disorders) | 1 | 0
Poisoning (Investigations) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Follicle centre lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Blood and lymphatic system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=70) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 2 | 4
Influenza (Infections and infestations) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Headache (Nervous system disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.